CLINICAL TRIAL: NCT02899234
Title: Acute Health Effects of Exposure to Active E-cigarette Inhalation in Healthy Volunteers
Brief Title: Acute Cardiorespiratory Effects of E-cigarette Inhalation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jenny Bosson, MD, PhD, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Umu-104-31
Record Dates: First submitted 2016-09-08; First posted 2016-09-14 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Nicotine; Electronic Cigarette
MeSH Terms: conditions — Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine-free e-cigarette (Active Comparator): Subjects will actively inhale nicotine-free vapor prior to blood samples and various non-invasive cardiopulmonary tests.
  Interventions: Other: E-cigarette
- Nicotine e-cigarette (Active Comparator): Subjects will actively inhale nicotine containing vapor prior to blood samples and various non-invasive cardiopulmonary tests.
  Interventions: Other: E-cigarette

INTERVENTIONS:
Other: E-cigarette — A third generation e-cigarette device will be used with pre-determined temperature, voltage and wattage settings.

SUMMARY:
According to the World Health Organization cigarette smoking is today one of the leading single causes of preventable death and morbidity. The electronic cigarette (e-cigarette) has been marketed as a safer alternative to conventional cigarettes, and its global sales continue to grow exponentially each year. Despite growing e-cigarette use, scientific data on health effects are insufficient in some respects and completely lacking in others. Therefore the current study is designed to investigate the effects of active e-cigarette inhalation on the cardiovascular and respiratory systems.

DETAILED DESCRIPTION:
It is estimated that 6 million people worldwide lose their lives due to tobacco use yearly. On average, cigarette smokers are estimated to die 10 years earlier than non-smokers. Ischemic heart disease, chronic obstructive pulmonary disease, stroke, respiratory illness, lung cancer and other cancers have all been linked to tobacco use. In recent years the electronic cigarette (e-cigarette) has been introduced to the market as an alternative to traditional cigarette smoking. E-cigarettes have been aggressively marketed as a cheaper, healthier, cleaner alternative to smoking in both advertising and media outlets, primarily targeting women and adolescents. With limited knowledge of e-cigarette vaping health effects in humans it has been challenging for governments and health officials to give advice and regulate the use of this novel product.

In the current study investigators aim to investigate acute cardiovascular and respiratory effects after active inhalation of e-cigarette in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent/sporadic cigarette smoking
* Normal clinical examination
* Normal EKG
* Normal blood tests
* Normal lung function

Exclusion Criteria:

* Cardiovascular disease
* Respiratory disease
* Systemic or chronic disorders or disease
* Symptoms of infection or inflammation within 2 weeks of the study
* BMI≥30
* Pregnancy
* Current habitual cigarette smokers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | 1 day
  Pulse wave analysis (PWA), pulse wave velocity (PWV). Expressed as Pulse wave velocity (m/s) och augmentation index adjusted for pulse 75 (%).

SECONDARY OUTCOMES:
Lung function | 1 day
  Assessed using spirometry testing.
Cardiovascular biomarkers | 1 day
  Blood samples are taken in order to assess cardiovascular biomarkers using microassay testing.
Impulse oscillometry | 1 day
  Non-invasive measurement by which to evaluate large and small airway resistance, and thereby also airflow obstruction.
Microcirculation assessment | 1 day
  Microcirculation assessment is performed using the GlycoCheck system. This measures the endothelial cell surface layer non-invasively by applying a clinical videomicroscope to the sublingual arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Bosson, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Dept of Medicine, Lung and Allergy section, University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided